CLINICAL TRIAL: NCT06022627
Title: EFFECT OF PRANAYAMA YOGA ON SYMPTOMS, FATIGUE AND RESPIRATORY PARAMETERS IN INDIVIDUALS WITH COPD
Brief Title: EFFECT OF PRANAYAMA YOGA ON COPD
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1707
Record Dates: First submitted 2023-07-23; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Asthma, Chronic Obstructive Pulmonary Disease (COPD), or Chronic Lung Disease (E.G., Chronic Bronchitis and Restrictive Lung Diseases Such as Asbestosis); The Effect of Yoga, Paranayama Yoga Practice on Respiratory Diseases
Keywords: Pranayama Yoga; COPD; Semptoms; Fatigue; Pulmonary functions
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Fatigue

STUDY DESIGN:
Intervention Model Description: 66 individuals with COPD included by randomization were divided into two groups as 33 (16 Stage I and 17 Stage II) study group and 33 (16 Stage I and 17 Stage II) control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayam Yoga Group (Experimental): It was planned to use a simple random sampling method among individuals who met the research inclusion criteria and agreed to participate voluntarily in the study. During randomization; Patients in the study and control groups will be determined using the random.org site. While the routine treatment of the patients in the study group continues, 20 minutes of pranayama yoga training will be given by the yoga instructor to the patient and his relatives, and it is planned that the patient will practice pranayama yoga, which is taught for 20 minutes every day for 21 days. Patients or their relatives will be called every morning by phone or video communication will be made online and pranayama yoga will be provided. In addition, a training booklet describing pranayama yoga exercises in detail, a training video and a 21-day checklist of doing yoga will be given to the patients. function test will be done and checklists will be taken back from patients.
  Interventions: Behavioral: Pranayama Yoga
- Non-Pranayama Yoga Group (No Intervention): The routine treatment of the control group will continue and any intervention will not be applied. After the data collection process of the study is completed, paranayama yoga training will be given to the patients in the control group and they will be advised to do it regularly for at least 21 days.

INTERVENTIONS:
Behavioral: Pranayama Yoga — Doing practice of paranayam yoga which including breathing exercises yoga-life energy
  Arms: Pranayam Yoga Group

SUMMARY:
The aim of the study In this study, pranayama yoga practices are the sub-dimensions of respiratory parameters, symptom and disease affection level, psychosocial adjustment and psychosocial adjustment in individuals with COPD. It was planned in a randomized controlled manner to examine the effects of healthcare compliance, professional environment, family environment, sexual relations, extended family relationships, social environment and psychological pressure. Pranayama yoga practices are aimed to reduce the frequency of symptoms and the level of disease exposure in individuals with COPD. Pranayama yoga practices are aimed to increase psychosocial adjustment in individuals with COPD. Pranayama yoga practices aim to increase compliance with health care, occupational, social and family environment, sexual and extended family relationships, and psychological pressure, which are the sub-dimensions of psychosocial adjustment in individuals with COPD. It is observed that all the yoga practices performed have improved the pulmonary functions of individuals with COPD, decrease the severity of symptoms, relieve inflammation, and increase muscle strength and physical performance. It was concluded that because of yoga increases awareness in patients, patients significantly reduce their level of depression and anxiety and adapt to social life. Yoga improves patients' quality of life by alleviating symptoms and increasing self-awareness. pranayama yoga practices are safe, home-applied, effective, cost-effective, complementary to drug therapy and can be performed during pulmonary rehabilitation for individuals with COPD (1-2) . The results of this study are important in guiding caregivers and healthcare professionals during the holistic care of COPD individuals and in pulmonary rehabilitation.

DETAILED DESCRIPTION:
Deep breathing exercises called pranayama yoga increase the oxygen and diffusion capacity of the alveolar in the lungs and facilitate gas exchange (1-3). Thus, tissue perfusion increases, more oxygen binds to hemoglobin and is transported (4-5).

Material and Method Purpose and Type of Study: This study was planned as a randomized controlled study to examine the effects of pranayama yoga practices on symptoms, fatigue and respiratory parameters in individuals with COPD.

Research Goals

1. Pranayama yoga practices are aimed to increase the FEV1, FVC, FV1/FVC … parameters of individuals with COPD.
2. Pranayama yoga practices are aimed at improving the symptom level of individuals with COPD.
3. Pranayama yoga practices are aimed at reducing fatigue levels in individuals with COPD.

Research Hypotheses H1: Pranayama yoga increases COPD respiratory parameters (FEV1, FVC, FV1/FVC, PEF, FEF AND VC) H2: Pranayama yoga reduces COPD symptom level H3: Pranayama yoga reduces COPD fatigue level

Patient selection and administration The study was conducted using simple random sampling method among individuals with COPD who met the inclusion criteria and voluntarily agreed to participate in the study. Patients GOLD, 2021 COPD classification, disease stages of the patients were determined and 66 patients with group B Stage I and Stage II COPD were included in the study. The patients included in the study were numbered by identifying the patients in the study and control groups using the random.org website. 66 individuals with COPD included by randomization were divided into two groups as 33 (16 Stage I and 17 Stage II) study group and 33 (16 Stage I and 17 Stage II) control group. According to the spirometric FEV 1 values of the patients in the study and control groups, 16 patients with Stage I and 17 Stage II COPD in each group were included in the study. While the routine treatment of the patients in the study group continued, 20 minutes of pranayama yoga training was given to the patient and his relatives by the yoga instructor (researcher), and it was planned that the patient would practice pranayama yoga, which was taught for 20 minutes a day for 21 days. In addition, patients will be given a training booklet detailing pranayama yoga exercises, a training video, and a 21-day checklist of practicing yoga. Patients or their relatives will be called every morning by phone or online communication will be established and pranayama yoga will be provided. After the application is over, the patients will be visited at the hospital or at their homes, and the re-interview form, COPD Assessment Test (CAT), COPD and Asthma Fatigue Scale (CAFS) will be filled and pulmonary function test will be performed and checklists will be taken back from the patients. The routine treatment of the control group will continue and no intervention will be applied. After the data collection process of the study is completed, paranayama yoga training will be given to the patients in the control group and they will be advised to do it regularly for at least 21 days.

Resources

1. Ranjita, R., Hankey, A., Nagendra, H. R., & Mohanty, S. (b2016). Yoga-based pulmonary rehabilitation for the management of dyspnea in coal miners with chronic obstructive pulmonary disease: a randomized controlled trial. Journal of Ayurveda and integrative medicine, 7(3), 158-166.
2. Soni, R., Munish, K., Singh, K. P., & Singh, S. (2012). Study of the effect of yoga training on diffusion capacity in chronic obstructive pulmonary disease patients: A controlled trial. International journal of yoga, 5(2), 123.
3. Zeng, Y., Jiang, F., Chen, Y., Chen, P., & Cai, S. (2018). Exercise assessments and trainings of pulmonary rehabilitation in COPD: a literature review. International journal of chronic obstructive pulmonary disease, 2013-2023.
4. Li, C., Liu, Y., Ji, Y., Xie, L., & Hou, Z. (2018). Efficacy of yoga training in chronic obstructive pulmonary disease patients: a systematic review and meta-analysis. Complementary therapies in clinical practice, 30, 33-37. doi: 10.1016/j.ctcp.2017.11.006
5. Pomidori, L., Campigotto, F., Amatya, T. M., Bernardi, L., & Cogo, A. (2009). Efficacy and tolerability of yoga breathing in patients with chronic obstructive pulmonary disease: a pilot study. Journal of cardiopulmonary rehabilitation and prevention, 29(2), 133-137. Available at: https://insights.ovid.com/pubmed?pmid=1930523.
6. Thokchom, S. K., Gulati, K., Ray, A., & Menon, B. K. (2018). Effects of yogic intervention on pulmonary functions and health status in patients of COPD and the possible mechanisms. Complementary Therapies in Clinical Practice, 33, 20-26. doi: 10.1016/j.ctcp.2018.07.008

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40-65
* To have been diagnosed with Stage I or Stage II COPD for at least six months
* Absence of any communication problem [decreased hearing, visual impairment, inability to understand/speak Turkish] that would prevent participation in the research,
* Least literate
* Do not have any mental or physical disability that would prevent them from practicing Pranayama Yoga.
* Not having done pranayama yoga before
* No tracheostomy
* Telephone communication is possible.
* The patients who accepted to participate in the study voluntarily constitute the sample of the study.

Exclusion Criteria:

* Being diagnosed with Stage III and Stage IV COPD,
* Patients under the age of 40 and not over the age of 65
* Individuals who are bored during the interview and give up on the interview will not be included in the study and their data will not be used.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2023-09-16 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
COPD Assesment Test (CAT) | 21 days
  Assesment Test

SECONDARY OUTCOMES:
SPIROMETER | 21 days
  MIR-Spirobank Portable Spirometer
Asthma Fatigue Scale (CAFS) | 21 days
  Assesment Test

CONTACTS AND LOCATIONS:
Locations (1):
- University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No